CLINICAL TRIAL: NCT00025467
Title: A Phase II Evaluation of Thalidomide (NSC #66847, IND 48832) in the Treatment of Recurrent of Persistent Endometrial Carcinoma
Brief Title: Thalidomide in Treating Patients With Recurrent or Persistent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02420; GOG-0229-B; U10CA027469 (NIH); CDR0000068964 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-10-11; First posted 2003-10-15 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Endometrial Adenoacanthoma; Endometrial Adenocarcinoma; Endometrial Adenosquamous Cell Carcinoma; Endometrial Clear Cell Carcinoma; Endometrial Papillary Serous Carcinoma; Recurrent Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Thalidomide

ARMS (1):
- Treatment (thalidomide) (Experimental): Patients receive oral thalidomide once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: thalidomide; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: thalidomide — Given orally
  Other Names: Kevadon; Synovir; THAL; Thalomid
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of thalidomide in treating patients who have recurrent or persistent endometrial cancer. Thalidomide may stop the growth of cancer by stopping blood flow to the tumor

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the antitumor cytostatic activity of thalidomide, in terms of 6-month progression-free survival, in patients with recurrent or persistent endometrial carcinoma.

II. Determine the nature and degree of toxicity of this drug in these patients. III. Determine the partial and complete response rates in patients treated with this drug.

IV. Determine the duration of progression-free and overall survival in patients treated with this drug.

V. Determine the effect of this drug on initial performance status and histological grade in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral thalidomide once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed endometrial carcinoma

  * Recurrent or persistent (refractory to curative therapy or established treatment)
  * No sarcomas
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques, including palpation, plain x-ray, CT scan, or MRI
  * At least 10 mm by spiral CT scan
* At least 1 target lesion outside the area of prior radiotherapy
* Received 1 prior chemotherapy regimen for endometrial carcinoma

  * Initial treatment may include high-dose therapy, consolidation, or extended therapy
  * No more than 1 additional cytotoxic regimen for recurrent or persistent disease
  * No non-cytotoxic chemotherapy for recurrent or persistent disease
* Ineligible for higher priority GOG protocols (any active GOG phase III protocol for the same patient population)
* No documented brain metastases since diagnosis of cancer

  * Patients with stable CNS deficits allowed provided there are no brain metastases, as confirmed by CT scan or MRI
* Performance status - GOG 0-2 if patient received 1 prior regimen
* Performance status - GOG 0-1 if patient received 2 prior regimens
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* Creatinine no greater than 1.5 times ULN
* Creatinine clearance greater than 60 mL/min
* Not pregnant
* Negative pregnancy test
* Fertile patients must use 2 methods of effective contraception for 4 weeks before, during, and for 4 weeks after study participation
* No active infection requiring antibiotics
* No sensory or motor neuropathy greater than grade 1
* No other invasive malignancy within the past 5 years except non-melanoma skin cancer
* No documented seizure disorders since diagnosis of cancer

  * Patients with a history of seizure disorders allowed provided that the seizures have been stable (i.e., no seizure within the past 12 months) while on an appropriately monitored treatment regimen
* At least 3 weeks since prior biologic or immunologic agents directed at malignancy
* No prior thalidomide
* See Disease Characteristics
* At least 3 weeks since prior chemotherapy directed at malignancy and recovered
* At least 1 week since prior hormonal therapy directed at malignancy
* Concurrent hormone replacement therapy allowed
* See Disease Characteristics
* At least 3 weeks since prior radiotherapy directed at malignancy and recovered
* No prior radiotherapy to more than 25% of marrow-bearing areas
* Recovered from prior surgery
* At least 3 weeks since any other prior therapy directed at malignancy
* No prior cancer therapy that would preclude study participation
* No concurrent bisphosphonates (e.g., zoledronate)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2001-09; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients alive and progression-free | 6 months
Frequency of adverse events assessed by CTC | Up to 6 years

SECONDARY OUTCOMES:
Progression-free survival | From study entry until disease progression, death, or date of last contact, assessed up to 6 years
Overall survival | From entry into the study to death or the date of last contact, assessed up to 6 years
Frequency of clinical response using the GOG RECIST criteria | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: D. Scott McMeekin, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States